CLINICAL TRIAL: NCT05548751
Title: Physiotherapy Assessment Based on the ICF Model in The Lesch-Nyhan Syndrome: Case Report
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, tuba kolaylı, Lecturer, Uskudar University
Other Study IDs: UskudarU.
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Lesch-Nyhan Syndrome
Keywords: case report; lesch-nyhan syndrome; genetic disorders
MeSH Terms: conditions — Lesch-Nyhan Syndrome; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lesch-Nyhan Syndrome (LNS) is a genetic disorder that results in a deficit in the hypoxanthine-guanine phosphoribosyltransferase (HPRT) enzyme, which affects purine metabolism. It is a genetic disorder that is carried by an X-linked recessive gene.

LNS has 3 typical symptoms. These are increased uric acid, neurological symptoms and behavioral disorders. Dystonia is often seen among its neurological manifestations. Signs of primidal and extraprimidal system can be seen.

It is very important to create the syndrome-specific physiotherapy program. In order to achieve this, evaluations based on the International Classification of Functioning, Disability and Health (ICF) model are valuable in terms of showing the right way in the management of the disease.

DETAILED DESCRIPTION:
Lesch-Nyhan Syndrome (LNS) is a genetic disorder that results in a deficit in the hypoxanthine-guanine phosphoribosyltransferase (HPRT) enzyme, which affects purine metabolism. It was described by Lesch and Nyhan in 1960. It is a genetic disorder that is carried by an X-linked recessive gene and is therefore predominantly seen in males.

LNS has 3 typical symptoms. These are increased uric acid, neurological symptoms and behavioral disorders. Self-harming behavior begins to appear from the age of 2. Dystonia is often seen among its neurological manifestations. Signs of primidal and extraprimidal system can be seen.

As developments in treatment methods continue in individuals with LNS, the expected life expectancy of these individuals is prolonged. However, these individuals require physiotherapy for symptoms specific to LNS.

Because of the developmental delay seen in babies with LNS, these babies may be diagnosed with cerebral palsy. It is very important to create the syndrome-specific physiotherapy program. In order to achieve this, evaluations based on the International Classification of Functioning, Disability and Health (ICF) model are valuable in terms of showing the right way in the management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Having lesch-nyhan syndrome

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A case who had the Lesch-Nyhan Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-09-26 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Demographic information form | 20 munites
  This form was prepared by the researchers to obtain the demographic data of the case in the study.
Gross Motor Function Measure (GMFM) | 45 minutes
  The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy, Down Syndrome and acquired brain damage.
Gross Motor Function Classification System (GMFCS) | 10 munites
  Gross Motor Function Classification System developed in 1997[1] to classify and describe the abilities of children and youth with cerebral palsy. Generally, the higher the level the poorer the functional ability of the child.
Modified Ashworth Scale | 10 minutes
  Modified Ashworth Scale (MAS) is used to assess spasticity. Modified Ashworth Scale (MAS) have been utilized in the following populations: stroke, spinal cord injury, cerebral palsy, traumatic brain injury, pediatric hypertonia and central nervous system lesions.
Functional Independence Measure (WeeFIM) | 10 minutes
  The WeeFIM II® System, a pediatric version of the Functional Independence Measure™ (FIM) System, documents and tracks functional performance in children and adolescents with acquired or congenital disabilities by measuring a child's need for assistance, in addition to the severity of disability.
The Pediatric Quality of Life Inventory (PedsQL) | 20 minutes
  The Pediatric Quality of Life Inventory (PedsQL) is a valid, practical, brief, standardized, generic, and self-reporting assessment tool to measure health-related quality of life HRQOL for pediatrics and adolescents, it can be carried by patients himself and their parents.The PedsQL 4.0 Generic Core Scales instrument is the last version of PedsQL contain 23-items, including formats for typically developing children and adolescents 2 to 18 years old.

CONTACTS AND LOCATIONS:
Overall Officials: tuba kolaylı, MSc., Principal Investigator — Uskudar University
Locations (1):
- Üsküdar Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided